CLINICAL TRIAL: NCT02544984
Title: The Anti-inflammatory Effect of Prophylactic Macrolides on Children With Chronic Lung Disease: a Double Blinded RCT
Brief Title: The Anti-inflammatory Effect of Prophylactic Macrolides on Children With Chronic Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ricardo A. Mosquera, Associate Professor of Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC-MS-14-0476
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Chronic Lung Disease
Keywords: prophylactic macrolides; RSV; chronic lung disease; respiratory infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): The control group will be provided with a placebo medication of similar taste, color, texture, and consistency as the study medication, and will be dispensed once a day on Monday, Wednesday, and Friday.
  Interventions: Drug: placebo
- azithromycin (Experimental): Patients will receive azithromycin at a dose of 5 mg/kg to be given once a day on Monday, Wednesday, and Friday. The dosage will be not be adjusted if a new weight is obtained during the trial period.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Patients will receive azithromycin at a dose of 5 mg/kg to be given once a day on Monday, Wednesday, and Friday. The dosage will not be adjusted if a new weight is obtained during the trial period.
  Arms: azithromycin
Drug: placebo — Patients will receive placebo at a dose of 5 mg/kg to be given once a day on Monday, Wednesday, and Friday. The dosage will not be adjusted if a new weight is obtained during the trial period.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if the prophylactic use of azithromycin will reduce the total number of days when unscheduled treatment is given outside of the home in a clinic, urgent care, emergency room or hospital setting between the respiratory illness season months (October 1-March 31) and subsequent 2 month follow-up (April and May)

DETAILED DESCRIPTION:
STUDY DESIGN AND METHODS

Overview:

This pilot randomized control trial (RCT) will enroll 92 children from 6 months to 6 years of age that have chronic lung disease (CLD) such as bronchopulmonary dysplasia during two pulmonary illness seasons. If the minimum number of patients (n=92) in Season 1 is achieved, we will then perform an interim analysis of the data. However, if recruitment does not reach 92patients during the first season we will continue to recruit in Season 2 (2016-2017). These children will all be patients who receive their primary medical care from either the High Risk Children Clinic or the similar High Risk Infant Clinic that cares for premature infants from discharge until age 2. Clinic records will be screened to determine eligibility. Patients that have parental consent will be given a baseline EKG, a nasal aspirate, an oscillometer reading (over 2 years of age only), and a six month supply of either the medication or the placebo at an initial study or office visit. The medication/placebo will be taken once a day for three days a week: Monday, Wednesday and Friday. The azithromycin medication will be dosed at 5 mg/kg/day. Adjustments in dosage amount will not be made during the 6 month trial. Any child that is eligible to receive Synagis will be given this every 28-30 days in clinic. Patients will be followed on a monthly basis and closely monitored for adverse reactions; this will occur by phone, in clinic during their regularly scheduled appointments, and/or during any necessary illness visits. Any children with adverse reactions will discontinue the medication, but will continue to be followed clinically. At any clinic visit in which a child presents with respiratory infections, including pneumonia, upper respiratory illness, bronchiolitis, etc., he/she will have an additional nasal aspirate and an oscillometer reading performed. At the completion of the six month treatment phase, each child will have a final EKG, final nasal aspirate and an oscillometer reading performed. Data will continue to be collected for the following twelve months, to monitor for respiratory illnesses.

Study Procedures:

Patients will be randomized by the REDCap statistical program in a double blind manner. Parents will then be provided with an entire 6 months of medication or placebo. Half of the patients will receive azithromycin at a dose of 5 mg/kg to be given once a day on Monday, Wednesday, and Friday. The dosage will not be adjusted during the trial period. The other half, the control group, will be provided with a placebo medication of similar taste, color, texture, and consistency, also to be taken once a day on Monday, Wednesday, and Friday. Both the study medication and the placebo will be dispensed from Corner Compounding Pharmacy, mixed with a fish-oil base to ensure a shelf life of more than six months, and flavored with citrus to improve palatability. Parents will be contacted monthly, either in clinic or by phone, to monitor for any adverse reactions, including rash, nausea, vomiting, diarrhea, or abdominal cramping. If a significant adverse reaction occurs, the medication will be discontinued. If an allergic reaction (such as rash or shortness of breath) is noted, the blind will be broken by Claudia Pedroza, the statistician, who is not involved with the project. This un-blinding will be done to note if it is an allergy to the medication.

After the initial appointment, at any face to face encounter (unscheduled sick visit or hospital admission/ER admission Monday through Friday) in which the patient presents with respiratory symptoms, the patient will be evaluated by the research coordinator or one of the co-investigators. Specifically, if a patient presents with the following symptoms: cough, wheeze, tachypnea, rhinorrhea, increased respiratory secretions, hypoxemia, and/or an increased oxygen requirement, an additional nasal aspirate sample and an oscillometry reading (for patients over 2 years of age) will be performed. These samples will also be stored in the office of Dr. Piedra. At the conclusion of the six month treatment phase, a final nasal aspirate sample, an oscillometer reading and EKG will be performed while the patients are in clinic for an office visit. There will be no expected study visits and no compensation will be provided for parents or patients.

Research Aims

Primary Aim: To determine if the prophylactic use of azithromycin will reduce the total number of days when one or more unscheduled medical encounters occur in a clinic, urgent care, emergency room (ER) or hospital setting during the 3-6 month study period and subsequent 2 months.

Secondary Aims:

1. To determine if the prophylactic use of azithromycin will reduce the total number of days when one or more unscheduled medical encounters occur for acute respiratory illness in a clinic, urgent care, ER or hospital setting during the 3-6 month study period and subsequent 2 months.
2. To determine if the administration of azithromycin will have a similar number of adverse side effects, or adverse events leading to unscheduled face-to-face clinic, urgent care, ER or hospital visit as compared to placebo during the 3-6 month study period and subsequent 2 months.
3. To determine if the prophylactic use of azithromycin will reduce healthcare costs during the 3-6 month study period and subsequent 2 months.

Exploratory Outcomes:

1. To determine if the prophylactic use of azithromycin will reduce the level of pro-inflammatory cytokines and additional biomarkers of disease including Lactate Dehydrogenase and Myeloid Peroxidase, by 10%.
2. To determine if the prophylactic use of azithromycin during the 3-6 months intervention will reduce the level of airway resistance of patients with CLD during respiratory illness from their baseline when compared to the placebo group as measured by an Airwave Oscillometry System
3. To determine if prophylactic use of azithromycin will reduce the total number of unscheduled face-to-face provider visits for respiratory related illness in a clinic, urgent care, emergency room or hospital setting in the 12 months after the intervention phase.

Data Analysis Plan:

Patients will be randomized to one of two different branches by the REDCap data base randomization program. This will be a double-blind placebo controlled study. Standard frequentist and Bayesian analyses will be performed using an intent-to-treat approach. Total hospital days, total ER visits (counting one day for each ER visit), and unscheduled clinic visits (counting one day for each visit) will be analyzed and related to treatment (Azithromycin vs Placebo), with logistic regression models and the treatment group as a covariate and random intercept to account for within patient correlation (due to multiple ED visits). To assess the probability of benefit, we will use Bayesian hierarchical models with interaction terms between treatment groups (Azithromycin vs Placebo) and predefined potential moderators. The groups will be stratified by synagis use and if they have a tracheostomy.

Sample size and power:

Based on data from our HRCC, we expect the control group to have 1.6 encounters per child-year (SD=1.66). Assuming a two-sided alpha = 0.05, a sample size of 92 (46/group) will have 80% power to detect a difference of 1 in the encounter rate between placebo and azithromycin groups (i.e., 1.6 vs 0.6 in encounter rate or 38% reduction). Power will be more limited for secondary outcomes but Bayesian analyses will provide an estimate of the probability of benefit in these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* children with a diagnosis of chronic lung disease (CLD) secondary to bronchopulmonary dysplasia (BPD) as defined by ATS.
* children who receive primary care at High Risk Infant Clinic or High Risk Children's Clinic

Exclusion Criteria:

* Children with Cystic Fibrosis or bronchiectasis
* Children with cardiac arrhythmias
* Children with cyanotic heart disease
* Children with colitis
* Children with a known Macrolide allergy
* Children taking medications known to interact with macrolides
* Children with short bowel syndrome
* Children with kidney or liver failure

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Mosquera, MD, Principal Investigator — University of Texas Medical School in Houston
Locations (1):
- High Risk Children's Clinic, Houston, Texas, United States

REFERENCES:
- [Derived] Mosquera RA, Yadav A, Romero-Lopez MDM, Magana-Ceballos IG, Hashmi SS, De Jesus Rojas W, Tellez ME, Riggs-Harpur K, Boricha FM, Reddy TS, John JL, Harris TS, Rodriguez-Martinez CE, Buendia J, McBeth KE, Jon CK, Stark JM, Colasurdo GN. The Effect of Chronic Azithromycin Use in Winter on Health Care Utilization for Children With Bronchopulmonary Dysplasia: A Double Blind Randomized Controlled Study (RCT). Pediatr Pulmonol. 2025 Oct;60(10):e71314. doi: 10.1002/ppul.71314. PMID 41090256
- [Derived] Mosquera RA, Gomez-Rubio AM, Harris T, Yadav A, McBeth K, Gonzales T, Jon C, Stark J, Avritscher E, Pedroza C, Smith K, Colasurdo G, Wootton S, Piedra P, Tyson JE, Samuels C. Anti-inflammatory effect of prophylactic macrolides on children with chronic lung disease: a protocol for a double-blinded randomised controlled trial. BMJ Open. 2016 Sep 16;6(9):e012060. doi: 10.1136/bmjopen-2016-012060. PMID 27638496

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The control group will be provided with a placebo medication of similar taste, color, texture, and consistency as the study medication. Patients will receive placebo at a dose of 5 mg/kg to be given once a day on Monday, Wednesday, and Friday. The dosage will not be adjusted if a new weight is obtained during the trial period.
- Azithromycin: The azithromycin group will receive azithromycin at a dose of 5 mg/kg to be given once a day on Monday, Wednesday, and Friday. The dosage will not be adjusted if a new weight is obtained during the trial period.
Period: Overall Study
Arm/Group | Placebo | Azithromycin
Started | 30 | 30
Completed | 28 | 28
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Azithromycin | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Count of Participants; unit: Participants]
  Age: 6 -24 months | 19 | 19 | 38
  Age: 24 months-72 months | 11 | 11 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 14 | 19 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 14 | 31
  Not Hispanic or Latino | 13 | 16 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 10 | 19
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 17 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Gestational Age [Count of Participants; unit: Participants]
  <28 weeks | 22 | 20 | 42
  28-31 weeks | 6 | 4 | 10
  32-36 weeks | 2 | 6 | 8
Number of Participants who Received Synagis Injection [Count of Participants; unit: Participants] | 14 | 16 | 30
Number of Patients with Tracheostomy [Count of Participants; unit: Participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Unscheduled Face-to-face Physician Visits (Clinic Visits, ER Visits, and Hospitalizations)
Description: Participants were observed for a minimum of 5 months and a maximum of 8 months, depending on when study enrollment occurred. Patients were recruited for this study on a rolling basis during the start of the winter season and then completed the intervention at the same time at the end of the winter season, which accounts for the variability in the amount of time participants were observed.
Time Frame: 5 to 8 months
Measure: Number; unit: visits
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 30 | 30
visits
  Unscheduled clinic visits for respiratory symptoms | 16 | 21
  Unscheduled clinic visits for other symptoms | 3 | 5
  Emergency room visits | 15 | 6
  Hospital admissions | 6 | 5
Statistical Analysis 1: Comparison: Placebo vs Azithromycin; The numbers of unscheduled clinic visits due to respiratory symptoms are compared; Test type: Superiority; p = 0.473, negative binomial model; negative binomial model adjusting for use of Synagis and tracheostomy
Statistical Analysis 2: Comparison: Placebo vs Azithromycin; Unscheduled clinic visits due to symptoms other than respiratory symptoms are compared; Test type: Superiority; p = 0.505, negative binomial model; negative binomial model adjusting for use of Synagis and tracheostomy
Statistical Analysis 3: Comparison: Placebo vs Azithromycin; Numbers of emergency room visits are compared; Test type: Superiority; p = 0.047, negative binomial model; negative binomial model adjusting for use of Synagis and tracheostomy
Statistical Analysis 4: Comparison: Placebo vs Azithromycin; Numbers of hospital admissions are compared; Test type: Superiority; p = 0.675, negative binomial model; negative binomial model adjusting for use of Synagis and tracheostomy

2. Secondary Outcome: Number of Adverse Events
Description: as for outcome 1
Time Frame: 5 to 8 months
Measure: Number; unit: adverse events
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 30 | 30
adverse events | 4 | 2
Statistical Analysis 1: Comparison: Placebo vs Azithromycin; Test type: Superiority; p = 0.435, negative binomial model; negative binomial model adjusting for use of Synagis and tracheostomy

3. Secondary Outcome: Healthcare Cost Associated With Respiratory Illness
Description: Participants were observed for a minimum of 5 months and a maximum of 8 months, depending on when study enrollment occurred. Patients were recruited for this study on a rolling basis during the start of the winter season and then completed the intervention at the same time during the end of the winter season, which accounts for the variability in the amount of time participants were observed.
Time Frame: 5 to 8 months
Population: Cost-effective analyses are only justified for interventions that are shown to be effective. Because the intervention at study (the macrolide azithromycin) showed no benefit and led to worse outcomes than those with usual care, an economic evaluation is not warranted and claims data was not collected.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Long Term Reduction in Respiratory Symptoms
Description: To determine if prophylactic use of azithromycin will reduce the total number of unscheduled face-to-face physician visit for respiratory related illness in a clinic, urgent care, emergency room or hospital setting during the following 12 months after the intervention.
Time Frame: 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Level of Airway Conductance
Description: To determine if prophylactic use of azithromycin will reduce level of airway resistance as measured by an Airwave Oscillometry System in subjects above 2 years of age, at the time of respiratory illnesses, during the 3-6 months intervention.
Time Frame: 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Level of Cytokines
Description: Using a standardize nasal wash procedure, respiratory samples will be collected at enrollment, at end of study, and during acute respiratory illness requiring face-to-face provider interaction. Children with a tracheostomy will have both a nasal wash sample and a tracheal aspirate sample collected. The respiratory samples will be stabilized with a universal transport media, processed and stored at -80 C for future testing. Testing will be performed for cytokines/chemokines; other biomarkers of disease such as LDH, MPO, and caspase; viral and bacterial respiratory pathogens; and microbiome.
Time Frame: 8 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 to 8 months - Participants were observed for a minimum of 5 months and a maximum of 8 months, depending on when study enrollment occurred. Patients were recruited for this study on a rolling basis during the start of the winter season and then completed the intervention at the same time during the end of the winter season, which accounts for the variability in the amount of time participants were observed.
Description: Parents were contacted biweekly, either in clinic or by phone, to monitor for any adverse reactions, including rash, nausea, vomiting, diarrhea, or abdominal cramping.
Arm/Group | Placebo | Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 3/28 | 2/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Azithromycin (N=28)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Lower than planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT02544984/Prot_SAP_000.pdf